CLINICAL TRIAL: NCT06589167
Title: Metabolic Dysfunction Among Egyptian Patients with Chronic HBV
Brief Title: Metabolic Syndrome and Fatty Liver Disease Among Egyptian Patients with Chronic HBV
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hadeer Abd EL-Sattar Mohammed, Resident doctor, Assiut University
Other Study IDs: Metabolic syndrome and NAFLD
Record Dates: First submitted 2024-08-09; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Metabolic Syndrome; Fatty Liver Disease
Keywords: Metabolic syndrome; Nonalcoholic fatty liver disease; hepatic steatosis
MeSH Terms: conditions — Metabolic Syndrome; Non-alcoholic Fatty Liver Disease; Fatty Liver

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
1. investigate the Prevalence of combined hepatic steatosis in patients with chronic HBV.
2. to evaluate clinical characteristics of chronic HBV patients combined with metabolic syndrome and hepatic steatosis

DETAILED DESCRIPTION:
* Hepatitis B virus (HBV) infection is a major global health problem, with an estimated 290 million infections worldwide. The estimated prevalence of HBV is about 1.4% in Egypt.
* Chronic hepatitis B describes a spectrum of disease usually characterised by the presence of detectable hepatitis B surface antigen (HbsAg) in the blood or serum for longer than 6 months. In some people, chronic hepatitis B is inactive and does not present significant health problems, but others may progress to liver fibrosis, cirrhosis and hepatocellular carcinoma (HCC). The progression of liver disease is associated with hepatitis B virus (HBV) DNA levels in the blood. The presence of HbeAg is typically associated with higher rates of viral replication and therefore increased infectivity.
* Metabolic syndrome is an accumulation of several disorders that includes central obesity, insulin resistance, hypertension, and atherogenic dyslipidemia .These disorders raise the risk of atherosclerotic cardiovascular disease, including myocardial infarction, cerebrovascular accidents, peripheral vascular diseases, insulin resistance, and type II diabetes mellitus.
* Obesity causes an estimated 4.7 million premature deaths per year. It was the fifth greatest preventable cause of death in 2017, accounting for 8.4% of all deaths worldwide. Egypt ranks 18th with the highest prevalence of obesity in the world.44.7% of adult women and 25.9% of adult men are living with obesity. Egypt's obesity prevalence is higher than the regional average of 20.8% for women and 9.2% for men.
* Nonalcoholic fatty liver disease (NAFLD) is a leading cause of liver disease worldwide.The estimated global prevalence of NAFLD among adults is 32% and is higher among males (40%) compared to females (26%) .NAFLD is defined as the presence of steatosis (i.e. more than 5% liver fat content) without coexisting etiologies of secondary steatosis such as alcohol abuse and drug-induced liver injury .
* Dysregulated fatty acid metabolism and lipotoxicity in NAFLD disease initiate activation of signaling pathways that enhance pro-inflammatory responses and disrupt hepatocyte cell homeostasis, promoting progression of NAFLD disease to NASH(Non Alcoholic Steatohepatitis), fibrosis and HCC and can affect HBV replication and immune encountering of HBV virus, which may further have impact on liver disease progression .Chronic HBV infection is suggested to have an influence on metabolic changes, which could lead to NAFLD development and the HBV-induced inflammatory responses and molecular pathways may constitute an aggravating factor in hepatic steatosis development. The altered immune homeostasis in both HBV infection and NAFLD could be associated with progression to HCC development.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 years.

Exclusion Criteria:

* Age below 18 years.
* Patients with combined HBV,HCV,HIV.
* Patients refused to contribute in this study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: total coverage of all patients with HBV aged 18-60 years,not combined with HCV or HIV.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-09-07 (Estimated); Primary Completion 2025-09-07 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
investigate the Prevalence of combined hepatic steatosis in patients with chronic HBV | baseline

SECONDARY OUTCOMES:
evaluate clinical characteristics of chronic HBV patients combined with metabolic syndrome and hepatic steatosis | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Hadeer Abd El-Sattar, Principal Investigator — Assiut University; Ghadaa Abdel rahman, Study Director — Assiut University; Bahaa Osman Taha, Study Director — Assiut University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mohammed H, Eshetie A, Melese D. Prevalence of hepatitis B virus and associated risk factors among adults patients at Dessie referral and Kemise general hospitals in northeastern Ethiopia. Health Sci Rep. 2022 May 22;5(3):e659. doi: 10.1002/hsr2.659. eCollection 2022 May. PMID 35620544
- [Background] Bhat M, Ghali P, Deschenes M, Wong P. Prevention and Management of Chronic Hepatitis B. Int J Prev Med. 2014 Dec;5(Suppl 3):S200-7. PMID 26622990
- [Background] National Clinical Guideline Centre (UK). Hepatitis B (Chronic): Diagnosis and Management of Chronic Hepatitis B in Children, Young People and Adults. London: National Institute for Health and Care Excellence (UK); 2013 Jun. Available from http://www.ncbi.nlm.nih.gov/books/NBK254250/ PMID 25473721
- [Background] Swarup S, Ahmed I, Grigorova Y, Zeltser R. Metabolic Syndrome. 2024 Mar 7. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK459248/ PMID 29083742
- [Background] Bovolini A, Garcia J, Andrade MA, Duarte JA. Metabolic Syndrome Pathophysiology and Predisposing Factors. Int J Sports Med. 2021 Mar;42(3):199-214. doi: 10.1055/a-1263-0898. Epub 2020 Oct 19. PMID 33075830
- [Background] Samson SL, Garber AJ. Metabolic syndrome. Endocrinol Metab Clin North Am. 2014 Mar;43(1):1-23. doi: 10.1016/j.ecl.2013.09.009. PMID 24582089
- [Background] Aboulghate M, Elaghoury A, Elebrashy I, Elkafrawy N, Elshishiney G, Abul-Magd E, Bassiouny E, Toaima D, Elezbawy B, Fasseeh A, Abaza S, Voko Z. The Burden of Obesity in Egypt. Front Public Health. 2021 Aug 27;9:718978. doi: 10.3389/fpubh.2021.718978. eCollection 2021. PMID 34513789
- [Background] Teng ML, Ng CH, Huang DQ, Chan KE, Tan DJ, Lim WH, Yang JD, Tan E, Muthiah MD. Global incidence and prevalence of nonalcoholic fatty liver disease. Clin Mol Hepatol. 2023 Feb;29(Suppl):S32-S42. doi: 10.3350/cmh.2022.0365. Epub 2022 Dec 14. PMID 36517002
- [Background] Tourkochristou E, Assimakopoulos SF, Thomopoulos K, Marangos M, Triantos C. NAFLD and HBV interplay - related mechanisms underlying liver disease progression. Front Immunol. 2022 Dec 5;13:965548. doi: 10.3389/fimmu.2022.965548. eCollection 2022. PMID 36544761
- [Background] Huang SC, Liu CJ. Chronic hepatitis B with concurrent metabolic dysfunction-associated fatty liver disease: Challenges and perspectives. Clin Mol Hepatol. 2023 Apr;29(2):320-331. doi: 10.3350/cmh.2022.0422. Epub 2023 Feb 1. PMID 36726053
- [Background] Dai YN, Xu CF, Pan HY, Chen MJ, Yu CH. Fatty liver is associated with significant liver inflammation and increases the burden of advanced fibrosis in chronic HBV infection. BMC Infect Dis. 2023 Sep 28;23(1):637. doi: 10.1186/s12879-023-08632-y. PMID 37770837
- [Background] Wong YJ, Nguyen VH, Yang HI, Li J, Le MH, Wu WJ, Han NX, Fong KY, Chen E, Wong C, Rui F, Xu X, Xue Q, Hu XY, Leow WQ, Goh GB, Cheung R, Wong G, Wong VW, Yu MW, Nguyen MH. Impact of fatty liver on long-term outcomes in chronic hepatitis B: a systematic review and matched analysis of individual patient data meta-analysis. Clin Mol Hepatol. 2023 Jul;29(3):705-720. doi: 10.3350/cmh.2023.0004. Epub 2023 May 8. PMID 37157776
- [Background] Liu L, Li H, Zhang Y, Zhang J, Cao Z. Hepatitis B virus infection combined with nonalcoholic fatty liver disease: Interaction and prognosis. Heliyon. 2023 Jan 20;9(1):e13113. doi: 10.1016/j.heliyon.2023.e13113. eCollection 2023 Jan. PMID 36747946